CLINICAL TRIAL: NCT07304778
Title: Evaluation of a Mobile AI-powered Decision Support System for Insulin Dosing and Glucose Prediction in Type 1 Diabetes: The glUCModel Clinical Trial Protocol
Acronym: glUCModel-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Bioinspired Intelligence SL (Unknown); Hospital de Toledo (Unknown)
Responsible Party: Principal Investigator, J. Ignacio Hidalgo, Full Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: glUCModel-HUT; PDC2022-133429-I00 (Other Grant/Funding Number: Agencia Estatal de Investigación -Ministerio de Ciencia, Innovación y Universidades-Gobierno de España); PID2021-125549OB-I00 (Other Grant/Funding Number: Agencia Estatal de Investigación -Ministerio de Ciencia, Innovación y Universidades-Gobierno de España); PID2024-158129OB-I00 (Other Grant/Funding Number: Agencia Estatal de Investigación -Ministerio de Ciencia, Innovación y Universidades-Gobierno de España)
Record Dates: First submitted 2025-11-30; First posted 2025-12-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2)
Keywords: Diabetes; Bolus recomendation; Artificial Intelligence
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants continue MDI therapy. The intervention group will additionally use the glUCModel app. CGM data from the final 2 weeks will be analyzed
  Interventions: Other: glUCModel app
- Control (No Intervention): Participants continue MDI therapy. CGM data from the final 2 weeks will be analyzed

INTERVENTIONS:
Other: glUCModel app — The intervention consists on using glUCModel, an application designed to help people with diabetes. It features a suite of artificial intelligence tools and statistical techniques for capturing and managing key information that people with diabetes need to track, as well as for predicting glucose values to aid users in informed decision-making.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of integrating predictive models into insulin therapy management via the user-centered glUCModel mobile app in People with Type 1 Diabetes Mellitus following Multiple Insulin Dosing therapy. Participants will be aged 18 to 65 years. The main questions it aims to answer are:

Does using the app improve glycaemic control, as measured by time in range? Does using the app reduce the number of episodes of hyperglycaemia and hypoglycaemia? Are the app's design and functionality adequate?

The study will comprise four phases:ses}):

* Screening phase: Informed consent, collection of sociodemographic and clinical data, and baseline Pittsburg, IFIS, and DTSQ questionnaires.
* Run-in phase: 2 weeks of standard care with CGM. Data will be used to generate personalized predictive models in the intervention group.
* Active treatment phase: Participants continue MDI therapy. The intervention group will additionally use the glUCModel mobile app. CGM data from the final 2 weeks will be analyzed.
* Evaluation and analysis phase: Participants will complete the uMARS, Pittsburgh, and DTSQ questionnaires. Statistical analysis and correlations among outcomes will be processed.

DETAILED DESCRIPTION:
Diabetes mellitus is a chronic, metabolic disorder characterized by impaired regulation of blood glucose, affecting more than 400 million people worldwide. Insulin, a hormone produced by the pancreas, facilitates the uptake of glucose into cells for energy production. In diabetes, either insufficient insulin is produced or the body cannot use it effectively, leading to persistent hyperglycemia. Over time, uncontrolled glucose levels can result in serious complications, including cardiovascular disease, neuropathy, retinopathy, and nephropathy. Effective management is therefore essential to prevent both acute and long-term adverse outcomes.

Two main forms of diabetes can be distinguished. Type 1 diabetes mellitus (T1DM) is an autoimmune condition in which pancreatic β-cells are destroyed, resulting in absolute insulin deficiency. It accounts for approximately 10% of all cases. Individuals with T1DM require lifelong insulin replacement therapy, typically delivered as multiple daily injections (MDI) or via an insulin pump. In contrast, type 2 diabetes mellitus (T2DM), the more prevalent form, is characterized primarily by insulin resistance. While insulin production is preserved in early stages, progressive dysfunction may ultimately necessitate pharmacological therapy, including insulin. Lifestyle interventions such as healthy diet and physical activity can delay or prevent T2DM onset and progression.

For individuals with diabetes, day-to-day self-management requires frequent glucose monitoring and insulin dose adjustments that must take into account meals, physical activity, stress, illness, and other factors. Capillary glucose meters and, more recently, continuous glucose monitoring systems (CGMs) have greatly improved access to real-time glucose data. However, interpreting these data and deciding on corrective actions remains challenging, and errors in insulin dosing can lead to hypoglycemia or persistent hyperglycemia. Both acute complications and the constant decision-making load contribute to reduced quality of life and treatment fatigue.

To support patients in these complex tasks, predictive models of glucose dynamics have been extensively investigated. Accurate prediction could enable early warnings of hypo- or hyperglycemia and assist in optimizing insulin therapy. The ultimate vision is the development of a fully automated ''artificial pancreas'' combining glucose sensing, insulin delivery, and robust prediction algorithms. Various machine learning (ML) approaches have been explored for glucose forecasting, including Genetic Programming , K-Nearest Neighbours , Grammatical Evolution, and, most prominently, Neural Networks. Among neural architectures, Long Short-Term Memory (LSTM) and other recurrent models have demonstrated strong performance for time-series data such as CGM traces, although convolutional and multilayer perceptron (MLP) networks have also been applied. Despite encouraging results, challenges remain in ensuring accuracy, robustness, and real-world usability across diverse patient populations.

Managing T1DM, particularly in patients using MDI, continues to pose a major challenge. While CGM and insulin pumps have improved outcomes, decisions about insulin dosing still depend heavily on patient intuition and experience, leaving room for error and variability. There is therefore a clear need for decision-support tools that combine predictive analytics with personalized recommendations to enhance safety, autonomy, and treatment adherence.

The glUCModel mobile application was developed to address this need. Since its early versions, it integrates proprietary, patented artificial intelligence models to provide real-time insulin recommendations, short-term glucose forecasts, and predictive alerts for hypo- and hyperglycemia. With a forecast horizon of up to two hours, the system aims to reduce glycemic variability and support timely corrective actions.

This protocol describes a randomized, open-label clinical study to evaluate the efficacy and safety of the glUCModel application in patients with T1DM using MDI therapy. The primary objective is to assess improvement in short-term glycemic control, measured by the percentage of time spent in target range (70-180 mg/dL). Secondary objectives include reductions in glycemic excursions, improved treatment satisfaction, and evaluation of usability and adherence in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c < 9%
* Currently following an MDI Bolus-Basal therapy.

  * Wearing CGMs connected to a mobile phone.
  * Spanish language proficiency.
  * Willingness to participate in the trial.
  * At least one year since the time of diabetes diagnosis.
  * Ability to use a mobile application like glUCModel.
  * Own a mobile phone running Android or iOS operating system.
  * Ability to follow a Portion-controlled diet for diabetes.
  * Educated to do an active management of insulin dosing

Exclusion Criteria:

* HbA1c < 9%.
* Not wearing CGMs.
* Non-Spanish language proficiency.
* Less than one year since the time of diabetes diagnosis
* Unable to use a mobile application like glUCModel
* Unable to follow a Portion-controlled diet for diabetes
* Unable to do an active management of insulin dosing.
* Diagnosed with a significant psychiatric disorder.
* Subjects in treatment with corticoids
* Patients who have required hospitalization or surgery in the last six months.
* Pregnancy or planning a pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | During the last 2 weeks of intervention
  Time in Range (TIR), defined as the percentage of time that interstitial glucose is between 70-180 mg/dL during the final 2 weeks of the intervention phase
Usability and adherence | Two weeks
  Patient-reported outcomes on usability and adherence through uMARS. The usability of the app will be evaluated using the Spanish Version of the User Version of the Mobile Application Rating Scale (uMARS). This scale provides a comprehensive and objective measure of app usability and consists of 20 items. Each item is rated on a 5-point scale, ranging from 1 (inadequate) to 5 (excellent).

SECONDARY OUTCOMES:
Frequency of Level 1 hypoglycemia | During the last 2 weeks of intervention
  Frequency in minutes of Level 1 hypoglycemia (40 ≤ CGM glucose < 55).
Frequency of Level 2 hypoglycemias | During the last 2 weeks of intervention
  Frequency in minutes of Level 2 hypoglycemia (55 ≤ interstitial glucose ≤ 70)
Frequency of Level 1 hyperglycemias | During the last 2 weeks of intervention
  Frequency in minutes of Level 1 hyperglycemia (180 ≤ CGM glucose ≤ 240).
Frequency of Level 2 hyperglycemias | During the last 2 weeks of the intervention
  Frequency in minutes of Level 2 hyperglycemia (241 ≤ interstitial glucose ≤ 400).
Duration of Level 1 hypoglycemias | During the last 2 weeks of intervention
  Average Duration in minutes of Level 1 hypoglycemia (40 ≤ CGM glucose < 55)
Duration of Level 2 hypoglycemia | During the last 2 weeks of intervention
  Average duration in minutes of Level 2 hypoglycemia (55 ≤ interstitial glucose ≤ 70).
Duration of Level 1 hyperglycemias | During the last 2 weeks of intervention
  Average duration in minutes of Level 1 hyperglycemia (180 ≤ CGM glucose ≤ 240).
Duration of Level 2 hyperglycemias | During the last 2 weeks of the intervention
  Average duration in minutes of Level 2 hyperglycemia (241 ≤ interstitial glucose ≤ 400).
Glycemic coefficient of variation | During the last 2 weeks of intervention
  Coefficient of Variation (CV) is calculated using the mean and the standard deviation of the glucose values. Coefficient of Variation (CV) is calculated by dividing the Standard Deviation by the mean of the glucose values.
Glycemic variability | During the last 2 weeks of intervention
  Glycemic variability is computed as the standard deviation. Standard Deviation (SD) is measured as the dispersion of glucose values from the average.
Accepted Recommendations | During the last 2 weeks of intervention
  Percentage of insulin recommendations accepted and applied by the user from the total number of recommendations requested.
Quality of predictions | During the last 2 weeks of intervention
  Quality of predictions measured using the Parkes Errod Grid analysis.
Treatment satisfaction | last 2 weeks of the intervention
  Treatment satisfaction using the Diabetes Treatment Satisfaction Questionnaire (DTSQ)

OTHER OUTCOMES:
Sleep Quality before the intervention | The day of the start of the intervention
  We will evaluate Sleep Quality before and after the intervention. The Pittsburg Sleep Quality Index (PSQI) will be used. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties. https://www.sleep.pitt.edu/psqi
Sleep Quality after the intervention | Two weeks after the day of the end of the intervention
  We will evaluate Sleep Quality before and after the intervention. The Pittsburg Sleep Quality Index (PSQI) will be used. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties. https://www.sleep.pitt.edu/psqi

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad Complutense de Madrid, Madrid, Madrid
  - Hospital Universitario de Toledo, Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
It depends on the autorization of the University